CLINICAL TRIAL: NCT07407270
Title: The Effects of Bilateral and Unilateral Perceptual-Motor Exercises on Manual Dexterity and Visuospatial Memory in Children With Nonverbal Learning Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allameh Tabatabai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Allameh Tabataba'i University
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-verbal Learning Disorder
Keywords: Perceptual-Motor exercise; Bilateral; Unilateral; Manual Dexterity; Visuospatial Memory; Non-verbal Learning Disorder
MeSH Terms: interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unilateral 1 - Free play activities followed by intervention (Other): Five participants of Unilateral main group, receive free-play and non-interventional activities during the first phase, followed by unilateral perceptual-motor exercises in the second phase of the experiment. This arm investigates the effects of Unilateral training and treatment order on manual dexterity and visuospatial memory in NVLD children.
  Interventions: Behavioral: Free-play activities followed by unilateral perceptual-motor (PM) training intervention
- Unilateral 2 - Unilateral interventional activities followed by free play (Other): Five participants of Unilateral main group, receive unilateral interventional activities during the first phase, followed by non-interventional and free-play activities in the second phase. This arm investigates the effects of Unilateral training and treatment order on manual dexterity and visuospatial memory in NVLD children.
  Interventions: Behavioral: Unilateral perceptual-motor (PM) training intervention followed by free-play activities
- Bilateral 1 - Free play activities followed by intervention (Other): Five participants of Bilateral main group, receive free-play and non-interventional activities during the first phase, followed by bilateral perceptual-motor exercises in the second phase of the experiment. This arm investigates the effects of Bilateral training and treatment order on manual dexterity and visuospatial memory in NVLD children.
  Interventions: Behavioral: Free play non-interventional exercises in first phase followed by bilateral interventional exercises
- Bilateral 2 - interventional activities followed by free play (Other): Five participants of Bilateral main group, receive bilateral interventional activities during the first phase, followed by non-interventional and free-play activities in the second phase. This arm investigates the effects of Bilateral training and treatment order on manual dexterity and visuospatial memory in NVLD children.
  Interventions: Behavioral: Bilateral perceptual-motor (PM) training intervention followed by free-play and non-interventional activities in Phase 2

INTERVENTIONS:
Behavioral: Unilateral perceptual-motor (PM) training intervention followed by free-play activities — The first 18 sessions (3 days per week) students took the unilateral (PM) exercise interventional training program, where they used only their left hand for participating in interventional training program. The second phase started after 18 sessions interventional exercises, with 6sessions (one session per week) of non-interventional , free-play, and self oriented activates.
  Arms: Unilateral 2 - Unilateral interventional activities followed by free play
Behavioral: Free-play activities followed by unilateral perceptual-motor (PM) training intervention — The first phase is 6sessions ( one session per week) of free-play and non-interventional activates followed by 18 sessions (three sessions per week) of interventional unilateral training program, where students have to use only their left hand for doing the assignments of protocol.
  Arms: Unilateral 1 - Free play activities followed by intervention
Behavioral: Bilateral perceptual-motor (PM) training intervention followed by free-play and non-interventional activities in Phase 2 — The first 18 sessions (three sessions per week) students took the bilateral (PM) exercise interventional training program, where they used their both hands for participating in interventional training exercises. The second phase started after 18 sessions interventional exercises, with 6sessions (one session per week) of non-interventional , free-play, and self oriented activates.
  Arms: Bilateral 2 - interventional activities followed by free play
Behavioral: Free play non-interventional exercises in first phase followed by bilateral interventional exercises — The first phase is 6sessions (one session per week) of free-play and non-interventional activates followed by 18 sessions (three sessions per week) of interventional bilateral training program, where students have to use their both hands for doing the assignments of protocol.
  Arms: Bilateral 1 - Free play activities followed by intervention

SUMMARY:
The goal of this semi-experimental study is to investigate whether bilateral (limbs of both sides of the body, such as left and right hands) perceptual-motor (PM) exercises and unilateral (limb of only one side of the body, such as only the left hand) PM exercises affect manual dexterity and visuospatial memory in children with nonverbal learning disorder (NVLD). Each type of perceptual-motor exercise (bilateral vs. unilateral) is delivered in two different ways. Within each method, free-play and non-interventional activities are scheduled at different times (e.g., at the beginning vs. the end of the intervention phase). The main questions this study aims to address are:

1. Which type of perceptual-motor (PM) exercise-bilateral or unilateral-is more effective in improving manual dexterity of left and right hands and visuospatial memory in children with nonverbal learning disorder (NVLD)?
2. Which training sequence in unilateral and bilateral groups-free-play and self-oriented activities followed by interventional exercises, or interventional exercises followed by free-play activities-has a greater impact on right and left hands manual dexterity and visuospatial memory scores in children with NVLD?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosing with Nonverbal Learning Disorder (NVLD) based on Wechsler Intelligence Scale for Children-Fifth Edition (WISC-V)

Exclusion Criteria:

* being left-handed

Ages: 7 Years to 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Right-hand Manual Dexterity | From enrollment to the end of treatment in each group at 12 weeks
  Pre-test scores are obtained using the Box and Blocks Test (BBT) to assess right hand manual dexterity scores before the start of the experiment. After 24 sessions, when participants have completed both the interventional and non-interventional training programs in each group (e.g., unilateral and bilateral training groups), the BBT is administered again to evaluate improvements in manual dexterity scores. Comparisons of pre-test and post-test scores within each subgroup are used to assess the effects of treatment type (unilateral vs. bilateral) and treatment order (interventional exercises in the first phase vs. non-interventional activities in the first phase) on right hand manual dexterity.
Left-hand Manual Dexterity | From enrollment to the end of treatment at 12 weeks.
  Pre-test scores are obtained using the Box and Blocks Test (BBT) to assess left hand manual dexterity scores before the start of the experiment. After 24 sessions, when participants have completed both the interventional and non-interventional training programs in each group (e.g., unilateral and bilateral training groups), the BBT is administered again to evaluate improvements in manual dexterity scores. Comparisons of pre-test and post-test scores within each subgroup are used to assess the effects of treatment type (unilateral vs. bilateral) and treatment order (interventional exercises in the first phase vs. non-interventional activities in the first phase) on left hand manual dexterity.
Visuospatial memory | From enrollment to the end of treatment at 12weeks
  Pre-test scores are obtained using the Chorsi Block Test (CBT) to assess visuospatial memory before the start of the experiment. After 24 sessions, when participants have completed both the interventional and non-interventional training programs in each group (e.g., unilateral and bilateral training groups), the CBT is administered again to evaluate progress in visuospatial memory. The comparison of pre-test and post-test scores within each subgroup allows assessment based on treatment type (unilateral vs. bilateral) and treatment order (interventional exercises in the first phase vs. non-interventional activities in the first phase) on visual spatial memory in NVLD children.

CONTACTS AND LOCATIONS:
Locations (1):
- Valiasr Girls' Primary School, Isfahan, Isfahan, Iran